CLINICAL TRIAL: NCT05217030
Title: Efficacy of Animal Assisted Therapy in the Treatment of Patients With Traumatic Brain Injury (AAT/TBI)
Brief Title: Efficacy of Animal Assisted Therapy in the Treatment of Patients With Traumatic Brain Injury
Acronym: AAT/TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Principal Investigator, Leslie Horton, RN, CCRN-K, Animal Assisted Care Coordinator, Inova Health Care Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1216
Record Dates: First submitted 2022-01-06; First posted 2022-02-01 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Traumatic Brain Injury
Keywords: Critical Care; TBI; Animal Assisted Therapy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Two groups of patients had comparison of measurements-one group received AAT; one group did not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal Assisted Therapy (Experimental): This group of patients with traumatic brain injury received AAT throughout the acute care hospitalization
  Interventions: Other: Animal assisted therapy
- Control (No Intervention): This group of patients with traumatic brain injury did not receive AAT throughout the acute care hospitalization

INTERVENTIONS:
Other: Animal assisted therapy — Patients in AAT group had handler place dog on bed and patient's hand was placed on dog. Bedside RN measured GCS, RLAS, LoCmds before and after intervention
  Other Names: AAT
  Arms: Animal Assisted Therapy

SUMMARY:
Patients admitted to the ED with moderate to severe traumatic brain injury defined by GCS less than or equal to 10 and confirmed by head CT scan or MRI were randomized into 2 groups: one receiving animal assisted therapy (AAT) and one not receiving animal assisted therapy. Efficacy of AAT was measured by patient's progression in the Glasgow Coma Scale (GCS), Rancho Los Amigos Scale (RLAS), and ability to follow multi-step commands (LoCmds).

DETAILED DESCRIPTION:
In this Level 3 prospective, randomized case control basic research study, investigators compared 2 groups, randomly assigned: patients receiving AAT during their hospital stay and those patients receiving usual care. Investigators recruited adult patients admitted to the TICU with a severe or moderate TBI; patients' legally authorized representatives provided consent for patients to be randomized into an intervention or control group. Patients were randomized to the intervention or control group in a 1:1 ratio; the randomization schedule was generated in advance by the study biostatistician utilizing a permuted block method with block sizes of 2 or 4. Study subjects' assigned groups were indicated on paper in a sealed envelope that was opened by the researchers upon receipt of signed informed consent form.

Investigators hypothesized the subjects in the intervention group would achieve higher elevation in Glasgow Coma Scale (GCS), Ranchos Los Amigos Scale (RLAS), and ability to follow commands than those in the control group. GCS, RLAS, and Levels of Command (LOCmd) scores were recorded by the bedside nurse for enrolled patients within 24 hours of consent. LOCmds were determined by the number of commands a patient could follow without prompting in between the commands. Subjects unable to follow any commands scored "0"; those able to follow one command scored "1," and so on, up to 3 commands without prompting. Intervention patients then received AAT with a dog, followed by the collection of post-intervention scores. The bedside RN assisted the handler in placing the dog onto the patient's bed and the patient was informed the dog was present. The patient's hand was placed on the dog and then the patient was instructed to open eyes and/or follow commands. The bedside RN assessed and the recorded the patient's responses before and after each AAI. Control patients' second set of scores were recorded after a researcher sat in the room without engaging the patient. The bedside RN assessed and recorded the patient before and after each control intervention. AAT and control activities, with associated data collection,continued every Monday, Wednesday, and Friday following initial measurements. Subjects remained enrolled in the study through discharge, or until the subject was recorded at RLAS 7, or until hospitalized over 28 days. Patients discharged from the study, but remaining in the hospital, were able to continue receiving AAT.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Trauma ED with GCS < 10 due to Traumatic Brain Injury via head CT scan and/or head MRI
* Primary language is Spanish or English
* Free of Infection Precautions
* No canine allergies or fears
* Consent to Study Obtainable

Exclusion Criteria:

* Not meeting inclusion criteria (n=58)

  * Declined to participate (n=21)
  * No next of kin for consent (n=147)
  * Unsurvivable injury (n=83)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Glasgow Coma Scale | measuring the change before and after each intervention while in study until hospitalized for a period of 28 days or reached a level of rancho los amigos scale of 7
  standard measure in acute care for level of consciousness with scale of 3 -15 and 15 being the higher level of consciousness
Rancho Los Amigo Scale | measuring the change before and after each intervention while in study until hospitalized for a period of 28 days or reached a level of rancho los amigos scale of 7
  standard measure in acute and rehab care for level of consciousness, and for purposes of this study, were measured from 1 to 7 with 7 being reflective of the higher level of consciousness
Level of Commands | measuring the change before and after each intervention while in study until hospitalized for a period of 28 days or reached a level of rancho los amigos scale of 7
  ability to follow 3-step commands and is used for measure level of cognition with 0 being the lowest and 3 being the score that reflects higher level of consiousness

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Horton, RN, MBA, CCRN, Principal Investigator — Inova Health Systems
Locations (1):
- Inova Fairfax Medical Campus, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brain Trauma Foundation. (2021). It Can Happen Anywhere, Anytime, to Anyone. Retrieved July 2021, Brain_Trauma_Foundation.pdf: http://braintrauma.org
- [Background] Lo J, Chan L, Flynn S. A Systematic Review of the Incidence, Prevalence, Costs, and Activity and Work Limitations of Amputation, Osteoarthritis, Rheumatoid Arthritis, Back Pain, Multiple Sclerosis, Spinal Cord Injury, Stroke, and Traumatic Brain Injury in the United States: A 2019 Update. Arch Phys Med Rehabil. 2021 Jan;102(1):115-131. doi: 10.1016/j.apmr.2020.04.001. Epub 2020 Apr 24. PMID 32339483
- [Background] Javali RH, Krishnamoorthy, Patil A, Srinivasarangan M, Suraj, Sriharsha. Comparison of Injury Severity Score, New Injury Severity Score, Revised Trauma Score and Trauma and Injury Severity Score for Mortality Prediction in Elderly Trauma Patients. Indian J Crit Care Med. 2019 Feb;23(2):73-77. doi: 10.5005/jp-journals-10071-23120. PMID 31086450
- [Background] Murthy R, Bearman G, Brown S, Bryant K, Chinn R, Hewlett A, George BG, Goldstein EJ, Holzmann-Pazgal G, Rupp ME, Wiemken T, Weese JS, Weber DJ. Animals in healthcare facilities: recommendations to minimize potential risks. Infect Control Hosp Epidemiol. 2015 May;36(5):495-516. doi: 10.1017/ice.2015.15. No abstract available. PMID 25998315
- [Background] Pet Partners. Pet Partners. Retrieved from https://petpartners.org. 2021
- [Background] Osterhoudt, S. R. Animal Assisted Therapy: Improving Patient Outcomes in the ICU. Excelsior College, School of Nursing. 2018
- [Background] Tracy MF, Chlan L. Nonpharmacological interventions to manage common symptoms in patients receiving mechanical ventilation. Crit Care Nurse. 2011 Jun;31(3):19-28. doi: 10.4037/ccn2011653. PMID 21632591
- [Background] Hedrin, M. (2018, 2). Therapy Dogs May Unlock Health Benefits for Patients in Hospital ICUs. Retrieved August 2021, from John Hopkins University: https://hub.jhu.edu/2018/02/12/therapy-dogs-could-help-icu-patients-
- [Background] Abate SV, Zucconi M, Boxer BA. Impact of canine-assisted ambulation on hospitalized chronic heart failure patients' ambulation outcomes and satisfaction: a pilot study. J Cardiovasc Nurs. 2011 May-Jun;26(3):224-30. doi: 10.1097/JCN.0b013e3182010bd6. PMID 21263346
- [Background] Cole KM, Gawlinski A. Animal-assisted therapy: the human-animal bond. AACN Clin Issues. 2000 Feb;11(1):139-49. doi: 10.1097/00044067-200002000-00015. PMID 11040560
- [Background] Aldaghlas, Tayseer. Burke, Christine. Chang, Yung-Fu. Horton, Leslie. Rizzo, Anne. Richmond, Robyn. Schmidt, Keilla. To Pet or Not: Canine Assisted Therapy and the Risk of Clostridium Difficile. International Conference on Healthcare-Associated Infections. Atlanta, Ga: SHEA/APIC. March 19, 2010. https://shea.confex.com/shea/2010/webprogram/Paper2497.html

DOCUMENTS (1):
  • Study Protocol (2014-06-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05217030/Prot_000.pdf